CLINICAL TRIAL: NCT01865201
Title: Effect of Edaravone on Radiation-induced Temporal Lobe Necrosis in Patients With Nasopharyngeal Carcinoma After Radiotherapy
Brief Title: Effect of Edaravone on Radiation-induced Temporal Lobe Necrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009001
Record Dates: First submitted 2013-05-26; First posted 2013-05-30 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Nasopharyngeal Carcinoma; Brain Necrosis
Keywords: Radiotherapy; Radiation-induced brain necrosis; Edaravone; Effectiveness; Safety
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Edaravone; Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Edaravone group (Experimental): Edaravone was used at a dose of 30mg,intravenously, twice per day, for 14 days. All patients also received common fundamental management, which was as follows: ①Methylprednisolone, administered by intravenous infusion at a 500mg daily for 3 consecutive days and then gradually tailed off in 30 days with administration of oral prednisolone. ②Dehydration drugs.
  Interventions: Drug: Edaravone
- Control group (Experimental): All patients in this group received common fundamental management, which was as follows: ①Methylprednisolone, administered by intravenous infusion at a 500mg daily for 3 consecutive days and then gradually tailed off in 30 days with administration of oral prednisolone. ②Dehydration drugs.
  Interventions: Other: Common fundamental management

INTERVENTIONS:
Drug: Edaravone — Be used at a dose of 30mg, intravenously, twice per day, for 14 days.
  Other Names: 3-Methyl-1-phenyl-2-pyrazolin-5-one
  Arms: Edaravone group
Other: Common fundamental management — common fundamental management, which was as follows: ①Methylprednisolone, administered by intravenous infusion at a 500mg daily for 3 consecutive days and then gradually tailed off in 30 days with administration of oral prednisolone. ②Dehydration drugs.
  Other Names: Methlprednisolone; Mannitol
  Arms: Control group

SUMMARY:
It is hypothesized that excessive generation of free radicals involves in the pathogenesis of radiation-induced brain necrosis. This study therefore evaluated the effect of free radical scavenger, edaravone, on radiation-induced temporal lobe necrosis (TLN) in patients with nasopharyngeal carcinoma (NPC) after radiotherapy.

DETAILED DESCRIPTION:
Radiation-induced temporal lobe necrosis (TLN) is the most serious sequelae of radiotherapy and impairs the patients' quality of life profoundly. Steroid is one of the conventional treatment methods for TLN. However, its response rate was still not so satisfactory (about 30%-35%).The mechanism of TLN is under exploring and not completely understood. It has been proposed recently that chronic oxidative stress and inflammation involve in the pathogenesis of radiation-induced late normal tissue injury.

Edaravone(3-methyl-1-phenyl-2-pyrazolin-5-one), which is proved to be an excellent free radical scavenger, has been applied to a wide range of oxidative stress-related diseases.Thus, it may exert a therapeutic effect on radiation-induced temporal lobe necrosis. To support this hypothesis, the investigators carried out a randomized study of combining edaravone with common fundamental management versus common fundamental therapy in patients with TLN, and analyzed the Late Effects of Normal Tissues -Subjective, Objective, Management, Analytic (LENT/SOMA) scale before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* ①Patients must have received radiation therapy for histologically confirmed nasopharyngeal carcinoma.

  * Prior irradiation >/= 6 months prior to study entry.

    * Radiographic evidence to support the diagnosis of radiation-induced temporal lobe necrosis without tumor recurrence(15).

      * Age>/= 18 years.

        * No evidence of very high intracranial pressure that suggests brain hernia and need surgery.

          * Fertile women who are willing to take contraception during the trial.

            * Routine laboratory studies with bilirubin </=2 * upper limits of normal (ULN), aspartate aminotransferase (AST or SGOT) < 2 * ULN, creatinine <1.5 * ULN, red-cell count >/= 4,000 per cubic millimeter; white-cell count >/=1500 per cubic millimeter, platelets >/= 75,000 per cubic millimeter; Hb >/=9.0. prothrombin time(PT), activated partial thromboplastin time(APTT),international normalized ratio(INR) in a normal range.

              * Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* ①Tumor recurrence or metastases.

  * Diseases of central nervous system, such as cerebral vascular events, inflammatory, degenerative disease, and significant cardiovascular diseases.

    * Severe systemic diseases.

      * History of anaphylactic response to edaravone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-03; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The change of the maximum area of the necrosis lesion on MRI three months after treatment | At three months after treatment
  The radiographic response was assessed by difference between MRI pretreatment and post-treatment, which included T1-weighted gadolinium contrast-enhanced and T2-weighted image. The maximum area measurement of the radiation necrosis lesions were recorded (the product of the longest trans diameter and its longest perpendicular). And the change of the maximum area of the necrosis lesion on MRI three months after treatment was used as the secondary end point.

SECONDARY OUTCOMES:
The change in LENT/SOMA scale scores at three months after treatment from base line | Three months after treatment
  Clinical symptoms and signs were evaluated by Late Effects of Normal Tissues -Subjective, Objective, Management, Analytic (LENT/SOMA) scale(16) before drug administration and three months after treatment. Subjective domain contains five items: headache, somnolence, intellectual deficit, functional competence, and memory. Objective domain contains four items: neurologic deficit, cognitive functions, mood & personality changes, and seizures. And Analytic domain includes neuropsychologic and radiologic assessments. Each domain scores from 0 to 4. The summary of each domain represents the final score of LENT/SOMA scale. The primary end point was the change in LENT/SOMA scale scores at three months after treatment from base line.

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, M.D.,PhD., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Tang Y, Rong X, Hu W, Li G, Yang X, Yang J, Xu P, Luo J. Effect of edaravone on radiation-induced brain necrosis in patients with nasopharyngeal carcinoma after radiotherapy: a randomized controlled trial. J Neurooncol. 2014 Nov;120(2):441-7. doi: 10.1007/s11060-014-1573-4. Epub 2014 Aug 21. PMID 25142813
- See also: The homepage of Sun Yat-sen Memorial Hospital, Sun Yat-sen University — http://www.syshospital.com/